CLINICAL TRIAL: NCT01011790
Title: Evaluation of a Biofeedback-assisted Meditation Program as a Stress Management Tool for Hospital Nurses: A Pilot Study
Brief Title: Evaluation of a Biofeedback-assisted Meditation Program as a Stress Management Tool for Hospital Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Wild Divine (Unknown)
Responsible Party: Principal Investigator, Brent A. Bauer, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-002094
Record Dates: First submitted 2009-11-09; First posted 2009-11-11 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Stress
Keywords: Healing Rhythms™; Meditation; Biofeedback; Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stress Management Tool (Experimental): All subjects will use the Healing Rhythms™ meditation program for 4 weeks.
  Interventions: Behavioral: Healing Rhythms™ Meditation Program

INTERVENTIONS:
Behavioral: Healing Rhythms™ Meditation Program — The Healing Rhythms™ meditation program was chosen as the intervention for this study because it has a long history of use in the consumer market, it provides a dual-mode biofeedback which allows users to visually see their progress, and it provides an attractive and engaging user interface which is enjoyable to use. This is a critical factor as the research cited documents the importance of adherence in achieving optimal outcomes.
  Other Names: Wild Devine

SUMMARY:
The purpose of this study is to assess a novel meditation program which is biofeedback reinforced (Healing Rhythms™) as a means to improving stress management in a population of nurses practicing in the hospital setting.

DETAILED DESCRIPTION:
Stress is a common problem with significant ramifications for health. This is especially true in the workplace and particularly true for nurses practicing in a hospital environment. A number of factors (e.g. an aging population, the obesity epidemic, patients presenting with multi-system diseases, etc.) have dramatically increased the demands on hospital nurses in the past decade. This increased stress has potential ramifications at a personal level (e.g. increased risk of ill health) as well as an institutional (e.g. higher staff turnover). Meditation has been shown to be an effective tool for stress management. A self-directed, computer-guided meditation training program that can be pursued independently may be particularly useful for hospital nurses where scheduling challenges may preclude the use of scheduled classes. Healing Rhythms™ is a computer program that teaches meditation and uses biofeedback (heart rate variability and galvanic skin response) to reinforce the training.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 18 years of age
* Subjects that have given consent to participate
* Subjects that have access to a home computer

Exclusion Criteria:

* Subjects who are currently engaged in a routine meditative practice

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Assess the efficacy of a novel meditation program on stress, anxiety and quality of life (QOL) in nurses practicing in the hospital. Compare the level of stress, anxiety and QOL before and after a 4 week training period utilizing Healing Rhythms™. | 4 Weeks

SECONDARY OUTCOMES:
Evaluate feasibility of integrating a novel meditation program into an overall stress management program for nurses practicing in the hospital. Report overall satisfaction and identify challenges with the experience of the meditation program. | 4 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Susanne M. Cutshall, R.N., C.N.S., Principal Investigator — Mayo Clinic; Brent A. Bauer, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Cutshall SM, Wentworth LJ, Wahner-Roedler DL, Vincent A, Schmidt JE, Loehrer LL, Cha SS, Bauer BA. Evaluation of a biofeedback-assisted meditation program as a stress management tool for hospital nurses: a pilot study. Explore (NY). 2011 Mar-Apr;7(2):110-2. doi: 10.1016/j.explore.2010.12.004. PMID 21397872